CLINICAL TRIAL: NCT05117008
Title: A Multicenter Phase II Study of Maintenance Belantamab Mafodotin (Blenrep®) After BCMA-Directed Chimeric Antigen Receptor T-cell Therapy in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Maintenance Belantamab Mafodotin (Blenrep®) After B-cell Maturation Antigen-Directed Chimeric Antigen Receptor T-cell Therapy in Patients With Relapsed and/or Refractory Multiple Myeloma
Acronym: EMBRACE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Meera Mohan, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00042276
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Refractory Multiple Myeloma; Relapse Multiple Myeloma
Keywords: CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- belantamab mafodotin (Experimental): Belantamab mafodotin is an intravenous drug.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered IV over approximately 30 minutes at the recommended dose of 2.5 mg/kg IV over 30 minutes on day 1 of every eight-week (+/- three days) cycle for a maximum of 12 cycles. Maintenance therapy with belantamab mafodotin will continue until progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or end of study (maximum of 12 cycles), whichever occurs first.
  Other Names: Blenrep

SUMMARY:
This is a multicenter phase II, open-label study evaluating the efficacy and safety of belantamab mafodotin maintenance in participants with relapsed and/or refractory multiple myeloma (RRMM) who have received commercially available anti-BCMA CAR-T-cell therapy. Subjects will be enrolled 60-130 days after chimeric antigen receptor T-cell therapy (CAR-T) and receive belantamab mafodotin as maintenance therapy. Each maintenance cycle will have a duration of 56 days (+/- three days) and belantamab mafodotin will be administered at a dose of 2.5 mg/kg IV on day 1 of each cycle.

DETAILED DESCRIPTION:
INTERVENTION DESCRIPTION:

Subjects will receive belantamab mafodotin as maintenance therapy. Belantamab mafodotin will be administered IV over approximately 30 minutes at the recommended dose of 2.5 mg/kg IV over 30 minutes on day 1 of every eight-week (+/- three days) cycle for a maximum of 12 cycles. Maintenance therapy with belantamab mafodotin will continue until progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or end of study (maximum of 12 cycles), whichever occurs first. Dose interruptions or reductions may be required to address potential drug-associated toxicities. The dose to be administered will be based on actual body weight calculated at baseline. However, if the change in body weight is greater than 10%, the dose will be recalculated based on the actual body weight at the time of dosing. The dose may be reduced to address toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of multiple myeloma with measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥200 mg/24 hour or involved serum-free light chain ≥10 mg/dL provided that the ratio of involved/uninvolved light chain is abnormal) prior to receiving CAR-T. Patients with no biochemically measurable disease before CAR-T may be enrolled if bidirectionally measurable plasmacytomas or bone marrow plasmacytomas >10% are present prior to CAR-T infusion (sites must explicitly identify these patients to the Medical College of Wisconsin Multisite Team upon enrollment, as only four of these patients will be permitted on study, after which no future patients will be permitted to be enrolled).
2. Received at least three prior therapies (including a PI, immunomodulatory drugs (IMiD), and anti-cluster of differentiation 38 antibody (anti-CD38 antibody) ) given before CAR-T, and has not progressed/relapsed after receiving CAR-T therapy.
3. Achieved at least stable disease (SD) to CAR-T therapy and remained progression free after anti-BCMA CAR-T administration until enrollment (this requirement is also necessary prior administration of first study drug).
4. Voluntary consent (per single Institutional Review Board (sIRB) requirements) must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
5. Age ≥ 18 years.
6. Life expectancy ≥ six months.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Creatinine clearance (CrCl) ≥ 30 mL/minute, either measured or calculated using a standard formula (e.g., Modification of Diet in Renal Disease (MDRD) Study equation; Cockcroft and Gault).
9. Adequate hepatic function evidenced by aspartate aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 x ULN, bilirubin ≤ 1.5 x upper limit of the normal range (ULN) (isolated bilirubin ≥1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
10. Adequate bone marrow function evidenced by hemoglobin ≥8 g/dL, platelets ≥75,000/mm3 (without transfusion of platelets in the prior seven days) and absolute neutrophil count ≥1,500/mm^3 (growth factors are allowed during screening, but not within seven days prior to obtaining this result).
11. Spot urine (albumin/creatinine ratio) < 500 mg/g (56 mg/mmol) OR urine dipstick negative/trace (if ≥ 1+ only eligible if confirmed < 500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void).
12. Patients with prior allotransplant more than one year prior to enrollment, with or without ongoing topical treatment for skin GVHD (without evidence of active GVHD) are eligible (refer to exclusion criteria).
13. Female participants:

    Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    Is not a woman of childbearing potential (WOCBP). OR Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the intervention period and for four months after the last dose of belantamab mafodotin and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

    • WOCBP must have a negative highly sensitive serum pregnancy test within 72 hours of dosing on cycle 1 day 1 (C1D1) and agree to use a highly effective method of contraception during the study and for four months after the last dose of belantamab mafodotin.
14. Male participants:

Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Male participants are eligible to participate if they agree to the following from the time of first dose of study until six months after the last dose of belantamab mafodotin to allow for clearance of any altered sperm:

Refrain from donating sperm.

AND either:

Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

OR

Must agree to use contraception/barrier as detailed below:

• Agree to use a male condom, even if they have undergone a successful vasectomy and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as described in when having sexual intercourse with a WOCBP (including pregnant females).

Exclusion Criteria:

1. Prior disease refractoriness to belantamab mafodotin (progression on or within 60 days of enrollment.) This requirement is also necessary prior administration of first study drug).
2. Prior use of belantamab mafodotin with discontinuation of therapy due to toxicity.
3. Patient was given BCMA CAR-T under expanded access protocol (EAP) for non-conforming product.
4. Any previous treatment-related adverse events higher than grade 1 at enrollment (except for alopecia and grade 2 neuropathy).
5. Acute active infection requiring treatment within 14 days of enrollment (this requirement is necessary also prior administration of first study drug).
6. Current or prior involvement of central nervous system by multiple myeloma.
7. Smoldering multiple myeloma or POEMS.
8. Pregnant or lactating females.
9. Major surgery within 30 days prior to enrollment (this requirement is necessary also prior administration of first study drug).
10. Human immunodeficiency virus infection.
11. Evidence of cardiovascular risk including any of the following:

    1. Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including second-degree (Mobitz Type II) or third-degree atrioventricular (AV) block.
    2. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three months of enrollment.
    3. Class III or IV heart failure as defined by the New York Heart Association functional classification system (NYHA, 1994)
    4. Uncontrolled hypertension.
12. Nonhematologic malignancy within the past three years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason score 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
13. Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
14. Participant must not have current corneal epithelial disease except mild changes in corneal epithelium.
15. Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
16. Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria.
17. Participant must not use contact lenses while participating in this study.
18. Participant must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding enrollment (this requirement is also necessary prior administration of first study drug).
19. Participant must not have had plasmapheresis within seven days prior to enrollment (this requirement is also necessary prior administration of first study drug).
20. Participant must not have received prior treatment with a monoclonal antibody within 30 days of enrollment (this requirement is also necessary prior administration of first study drug).
21. Participant must not have had major surgery ≤ four weeks prior to enrollment (this requirement is also necessary prior administration of first study drug).
22. Participant must not have any evidence of active mucosal or internal bleeding.
23. Participant must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
24. Participant must not have known HIV infection.
25. Participant must not have presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within three months prior to first dose of study treatment. Note: presence of hepatitis B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant.
26. Participant must not have positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within three months prior to first dose of study treatment.

    Note: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C RNA test is obtained.

    Note: Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
27. Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least two years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a two-year restriction.
28. Prior allogenic stem cell transplant within one year before enrollment, or current evidence of GvHD, or on systemic immunosuppressive therapy for GvHD at least six weeks before enrollment. Note - Participants who have undergone syngeneic transplant will be allowed, only if no history of GvHD
29. Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
30. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
31. Administration of live or live-attenuated vaccines are contraindicated 30 days prior to the first dose of study treatment. Killed or inactivated vaccines may be administered; however, the response to such vaccines cannot be predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meera Mohan, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Belantamab Mafodotin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With 12-month Progression-free Survival.
Description: The primary endpoint of the study is the 12-month progression-free survival (PFS) with time counted from the CAR-T infusion conditional on being alive and progression-free at day +90 post CAR-T. An event will be defined as documented progression or death for any cause, subjects without an event will be censored at the last date known to be alive without progression.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Belantamab Mafodotin
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin (N=1)
acquired torsion dystonia (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (2)
Blurred Vision, Right eye (Eye disorders) | 1 (1)
Cervical dystonia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Corn, Left plantat feet (Skin and subcutaneous tissue disorders) | 1 (1)
Corneal Stromal scar, both eyes (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Corneal toxicities (Eye disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Genital Herpes (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Infertility (Reproductive system and breast disorders) | 1 (1)
Knee pain (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fatigue (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT05117008/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT05117008/ICF_001.pdf